CLINICAL TRIAL: NCT04239053
Title: Measurement of Bupivacaine Level Following ESPB (Erector Spinae Plane Block ) as a Part of Multimodal Analgesia
Brief Title: Bupivacaine Levels After ESPB
Status: Completed | Type: Observational
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Onur Selvi, Associate professor, Maltepe University
Other Study IDs: 01.10.2019 no 2
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia; Bupivacaine Adverse Reaction
Keywords: Bupivacaine; Erector Spinae Plane Block
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ESPB block group: Patients receiving ESPB will be enrolled to this group.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Measuring the plasma concentration level of bupivacaine after applying ESPB

SUMMARY:
Erector Spinae Plane Block (ESPB) is a regional anesthesia technique that is used for as a part of multimodal analgesia. Bupivacaine is one of the local anesthetic drugs and it is applied for ESPB. In this study, it is aimed to examine its blood concentration following the application for ESPB regarding its adverse effects and pharmacokinetics.

DETAILED DESCRIPTION:
ESPB is prefered block technique for thoraco abdominal surgeries. Bupivacaine is a widely used drug for these kind blocks.The systemic absorption rate of bupivacaine depends on the dose administered, the route of administration, and the vascularization of the injection site. The highest plasma concentration is achieved in intercostal blocks due to its rapid absorption (4 mg / liter after 400 mg dose).

The lowest plasma concentrations are seen in subcutaneous administration in the abdominal region. Total plasma clearance of bupivacaine was 0.58 L / min, steady state distribution volume was 73 liters, the elimination half-life was 2.7 hours and the hepatic extraction rate was 0.40. The maximum applicable legal dose varies by country. While it is 150 mg in Sweden, it is administered up to 400 mg in 24 hours in Finland. Clearance of bupivacaine has been shown to be lower in uremic patients. Plasma concentrations of highly proteing binding drugs are significantly effected by low cardiac output. The pharmacokinetics of many local anesthetics are influenced by inadequate liver function due to changes in body fluids and circulation. However, it seems safe in single dose blocks in patients with hepatic dysfunction. CYP2D6 enzyme inhibitors such as propranolol and CYP3A4 inhibitors such as itraconazole can reduce the clearance of bupivacaine by up to 30%.

As the concentration of local anesthetics including bupivacaine increases in systemic circulation, signs and symptoms of cardiovascular central nervous systems appear. The doses of bupivacaine that produce cardiovascular toxicity / central nervous system toxicity are similar. Stopping the administration of local anesthetics when early signs of the central nervous system observed does not prevent cardiotoxicity. Therefore, measurement of plasma levels of the drug may be important.

The blood level of bupivacaine is not routinely measured. Bupivacaine When the arterial plasma concentration is above 1.5 /g / ml, dizziness may occur, peripheral paresthesia above 2.0 /g / ml, and convulsions above 4.0 /g / ml. Intramuscular administration of 1.3 ug/kg causes psychomotor impairment in motor vehicle use. Dose-dependent central nervous system adverse effects are monitored and patient-related adverse event information is recorded. In a study in which toxic effects were observed with bupivacaine, which included 11,080 patients, the number of systemic toxicities was found to be 15 and none of them had permanent sequelae.

There are no reports on plasma bupivacaine levels in patients undergoing ESPB.

ELIGIBILITY:
Incluson criteria:

1. ESPB block receivers for thoracoabdominal surgeries
2. Patients stratified according to ASA
3. Female and male patients who underwent routine invasive arterial monitoring for additional diseases.
4. Who approved informed consent

Exclusion criteria:

1. Patients difficult to communicate
2. Patients does not give consent
3. uncontrolled hypertension
4. Patients with the previous diagnosis of neurological and psychiatric diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are already decided to be involved in Thoracoabdominal surgery who are decided to use bupivacaine with Erector spinae plane block before surgery for postoperative analgesia
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Bupivacaine plasma concentration | 10 sampling in 720 minutes after application.
  Determining plasma bupivacaine level after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University Medical Faculty, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No